CLINICAL TRIAL: NCT00903968
Title: Phase I/II Trial of Combination Plerixafor (AMD3100) and Bortezomib in Relapsed or Relapsed/Refractory Multiple Myeloma
Brief Title: Combination Plerixafor (AMD3100)and Bortezomib in Relapsed or Relapsed/Refractory Multiple Myeloma
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: Brigham and Women's Hospital (Other); Genzyme, a Sanofi Company (Industry); Millennium Pharmaceuticals, Inc. (Industry)
Responsible Party: Principal Investigator, Irene Ghobrial, MD, Principal Investigator, Dana-Farber Cancer Institute
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 08-273
Record Dates: First submitted 2009-05-18; First posted 2009-05-19 (Estimated); Results first posted 2017-09-29 (Actual); Last update posted 2020-06-02 (Actual); Status verified 2020-05

CONDITIONS: Multiple Myeloma
Keywords: refractory; relapsed; bortezomib; AMD3100; plerixafor
MeSH Terms: conditions — Multiple Myeloma; Recurrence | interventions — plerixafor; Bortezomib; Dexamethasone; Calcium Dobesilate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (9):
- Phase I Dose Level 1 (Experimental): Phase I Dose Level 1 patients received plerixafor 160ug/kg by injection on days 1-6 and bortezomib 1.0 mg/m2 intravenously days 3, 6, 10, and 13 of each 21 day cycle until disease progression or unacceptable toxicity.
  Interventions: Drug: Plerixafor; Drug: bortezomib
- Phase I Dose Level 2 (Experimental): Phase I Dose Level 2 patients received plerixafor 160ug/kg by injection on days 1-6 and bortezomib 1.3 mg/m2 intravenously days 3, 6, 10, and 13 of each 21 day cycle until disease progression or unacceptable toxicity.
  Interventions: Drug: Plerixafor; Drug: bortezomib
- Phase I Dose Level 3 (Experimental): Phase I Dose Level 3 patients received plerixafor 240ug/kg by injection on days 1-6 and bortezomib 1.0 mg/m2 intravenously days 3, 6, 10, and 13 of each 21 day cycle until disease progression or unacceptable toxicity.
  Interventions: Drug: Plerixafor; Drug: bortezomib
- Phase I Dose Level 4 (Experimental): Phase I Dose Level 4 patients received plerixafor 240ug/kg by injection on days 1-6 and bortezomib 1.3 mg/m2 intravenously days 3, 6, 10, and 13 of each 21 day cycle until disease progression or unacceptable toxicity.
  Interventions: Drug: Plerixafor; Drug: bortezomib
- Phase I Dose Level 5 (Experimental): Phase I Dose Level 5 patients received plerixafor 320ug/kg by injection on days 1-6 and bortezomib 1.3 mg/m2 intravenously days 3, 6, 10, and 13 of each 21 day cycle until disease progression or unacceptable toxicity.
  Interventions: Drug: Plerixafor; Drug: bortezomib
- Phase I Dose Level 5B (Experimental): Phase I Dose Level 5B patients received plerixafor 320ug/kg by injection on days 1, 2, 3, 6, 10, and 13 and bortezomib 1.3 mg/m2 intravenously days 3, 6, 10, and 13 of each 21 day cycle until disease progression or unacceptable toxicity.
  Interventions: Drug: Plerixafor; Drug: bortezomib
- Phase I Dose Level 6 (Experimental): Phase I Dose Level 6 patients received plerixafor 400ug/kg by injection on days 1, 2, 3, 6, 10, and 13 and bortezomib 1.3 mg/m2 intravenously days 3, 6, 10, and 13 of each 21 day cycle until disease progression or unacceptable toxicity.
  Interventions: Drug: Plerixafor; Drug: bortezomib
- All Phase I Participants (Experimental): All Phase I participants received plerixafor by injection and bortezomib intravenously according to the established dose escalation schedule. Participants were treated until disease progression or unacceptable toxicity.
  Interventions: Drug: Plerixafor; Drug: bortezomib
- All Phase II Participants (Experimental): All Phase I participants received plerixafor 320ug/kg by injection on days 1, 2, 3, 6, 10, and 13, bortezomib 1.3 mg/m2 intravenously or subcutaneously days 3, 6, 10, and 13, and dexamethasone 40mg orally days 3, 6, 10, and 13 of each 21 day cycle during induction. In maintenance, participants received plerixafor, bortezomib, and dexamethasone days 1, 8, 15, and 22 of each 35 day cycle. Participants were treated until disease progression or unacceptable toxicity.
  Interventions: Drug: Plerixafor; Drug: bortezomib; Drug: Dexamethasone

INTERVENTIONS:
Drug: Plerixafor
  Other Names: AMD3100
Drug: bortezomib
  Other Names: velcade
Drug: Dexamethasone
  Other Names: Decadron
  Arms: All Phase II Participants

SUMMARY:
The purpose of this research study is to determine the safety of plerixafor and bortezomib, and the highest dose that can be given to people safely. Plerixafor appears to stop myeloma cells from attaching to bone marrow and has been used in other phase I studies for mobilization of stem cells for patients with myeloma and lymphoma. We have shown that the combination of plerixafor and bortezomib is very effective in killing myeloma cells in the laboratory more than the effect of each drug alone.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Must have received prior 1-5 therapies for their myeloma and have relapsed or refractory multiple myeloma. Prior therapy with bortezomib is allowed as long as they were not refractory to bortezomib
* Monoclonal protein serum of 1gm/dL or greater or monoclonal light chain in the urine protein electrophoresis of 200 mg/24 hours or greater, or measurable light chains by free light chain assay of 10 mg/dL or greater, or measurable plasmacytoma
* ECOG Performance Status 0, 1, or 2
* Laboratory values as outlined in the protocol

Exclusion Criteria:

* Uncontrolled infection
* Cytotoxic chemotherapy < 3 weeks, or biologic or targeted novel therapy < 2 weeks, or corticosteroids < 2 weeks prior to registration. Patients may be receiving chronic corticosteroids if they are being given for disorders other than myeloma
* Pregnant women
* Nursing women
* Men or women of child-bearing potential who are unwilling to employ adequate contraception
* Other concurrent chemotherapy, immunotherapy, radiotherapy, or any ancillary therapy considered investigational
* Known to be HIV positive
* Radiation therapy < 2 weeks prior to registration

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2009-06-01 (Actual); Primary Completion 2016-06 (Actual); Study Completion 2016-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Irene Ghobrial, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (5):
- United States (5):
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Cape Cod Hospital, Hyannis, Massachusetts
  - Milford Hospital, Milford, Massachusetts
  - Newton-Wellesley Hospital, Newton, Massachusetts
  - Cancer Treatment Centers of America (Eastern Regional Medical Center), Philadelphia, Pennsylvania

REFERENCES:
- [Derived] Ghobrial IM, Liu CJ, Zavidij O, Azab AK, Baz R, Laubach JP, Mishima Y, Armand P, Munshi NC, Basile F, Constantine M, Vredenburgh J, Boruchov A, Crilley P, Henrick PM, Hornburg KTV, Leblebjian H, Chuma S, Reyes K, Noonan K, Warren D, Schlossman R, Paba-Prada C, Anderson KC, Weller E, Trippa L, Shain K, Richardson PG. Phase I/II trial of the CXCR4 inhibitor plerixafor in combination with bortezomib as a chemosensitization strategy in relapsed/refractory multiple myeloma. Am J Hematol. 2019 Nov;94(11):1244-1253. doi: 10.1002/ajh.25627. Epub 2019 Oct 4. PMID 31456261

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants in the Phase I study enrolled from June 2009 - July 2011 and the Phase II study from May 2012 - March 2015.
Groups:
- All Phase II Participants: All Phase II participants received plerixafor 320ug/kg by injection on days 1, 2, 3, 6, 10, and 13, bortezomib 1.3 mg/m2 intravenously or subcutaneously days 3, 6, 10, and 13, and dexamethasone 40mg orally days 3, 6, 10, and 13 of each 21 day cycle during induction. In maintenance, participants received plerixafor, bortezomib, and dexamethasone days 1, 8, 15, and 22 of each 35 day cycle. Participants were treated until disease progression or unacceptable toxicity.
Period: Overall Study
Arm/Group | Phase I Dose Level 1 | Phase I Dose Level 2 | Phase I Dose Level 3 | Phase I Dose Level 4 | Phase I Dose Level 5 | Phase I Dose Level 5B | Phase I Dose Level 6 | All Phase II Participants
Started | 3 | 3 | 3 | 3 | 4 | 6 | 3 | 33
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 3 | 3 | 3 | 3 | 4 | 6 | 3 | 33
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 8
Not completed — DLT | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 1 | 0 | 1 | 1 | 0 | 4
Not completed — Non-Compliance | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Physician Decision | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Progressive Disease | 2 | 3 | 2 | 3 | 3 | 3 | 0 | 18
Not completed — Lack of Efficacy | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3

BASELINE CHARACTERISTICS:
Groups:
- All Phase I Particiapnts: All Phase I participants received plerixafor by injection and bortezomib intravenously according to the established dose escalation schedule. Participants were treated until disease progression or unacceptable toxicity.
- Total: Total of all reporting groups
Arm/Group | All Phase I Particiapnts | All Phase II Participants | Total
Number analyzed (Participants) | 25 | 33 | 58
Age, Continuous [Median (Full Range); unit: years] | 59 [43 to 85] | 63 [46 to 83] | 63 [43 to 85]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 9 | 20
  Male | 14 | 24 | 38
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1
  Not Hispanic or Latino | 25 | 30 | 55
  Unknown or Not Reported | 0 | 2 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 0 | 4 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 1 | 3
  White | 22 | 27 | 49
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 25 | 33 | 58

OUTCOME MEASURES:

1. Primary Outcome: Plerixafor Maximum Tolerated Dose (MTD) [Phase I]
Description: The MTD plerixafor in combination with bortezomib is determined by the number of patients who experience a dose limiting toxicity (DLT). See subsequent primary outcome measure for the DLT definition. The MTD is defined as highest dose level at which fewer than one-third of patients experience a DLT. The MTD was reached at dose level 5B. The maximum tolerated dose of plerixafor was given on days 1, 2, 3, 6, 10, 13 of 21 each cycle.
Time Frame: Participants were assessed every 3 weeks while on study; The observation period for MTD evaluation was the first 21 days of treatment.
Population: All Phase I participants who received at least one dose of the study drug were evaluable for MTD.
Measure: Number; unit: ug/kg
Arm/Group | All Phase I Particiapnts
Number analyzed (Participants) | 25
ug/kg | 320

2. Primary Outcome: Bortezomib Maximum Tolerated Dose (MTD) [Phase I]
Description: The MTD plerixafor in combination with bortezomib is determined by the number of patients who experience a dose limiting toxicity (DLT). See subsequent primary outcome measure for the DLT definition. The MTD is defined as highest dose level at which fewer than one-third of patients experience a DLT. The MTD was reached at dose level 5B. The maximum tolerated dose of bortezomib was given on days 3, 6, 10, 13 of 21 each cycle.
Time Frame: as for outcome 1
Population: All Phase I participants who received at least one dose of the study drug were evaluable for MTD.
Measure: Number; unit: mg/m2
Arm/Group | All Phase I Particiapnts
Number analyzed (Participants) | 25
mg/m2 | 1.3

3. Primary Outcome: Number of Participants With Dose Limiting Toxicity (DLT) [Phase I]
Description: A DLT was defined as (a) grade 3 or greater non-hematologic toxicity, considered by the investigator to be related to plerixafor or bortezomib, with the exception of nausea, vomiting or diarrhea unless receiving maximal medical therapy, (b) grade 4 hematologic toxicity defined as: thrombocytopenia with platelets <10,000 on more than one occasion within first cycle despite transfusion. Grade 4 neutropenia must occur for more than 5 days and/or result in neutropenic fever with elevated temperature (defined as > 101 degrees F). (c) inability to receive Day 1 dose for Cycle 2 due to toxicity. All adverse events were graded according to the CTEP Common Toxicity Criteria (CTCAE v.3.0).
Time Frame: as for outcome 1
Population: All Phase I participants who received at least one dose of the study drug were evaluable for DLT.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase I Dose Level 1 | Phase I Dose Level 2 | Phase I Dose Level 3 | Phase I Dose Level 4 | Phase I Dose Level 5 | Phase I Dose Level 5B | Phase I Dose Level 6
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 4 | 6 | 3
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 2

4. Primary Outcome: Response Rate of Plerixafor, Bortezomib, and Dexamethasone in Relapsed or Relapsed/ Refractory Multiple Myeloma (ORR) [Phase I and Phase II]
Description: Overall response was established based on International Myeloma Working Group (IMWG) criteria with 6 potential categories: Complete Response (CR) which is a complete disappearance of monoclonal paraprotein based on negative immunofixation on the serum M-component and urine M-component and no evidence of myeloma in bone marrow, Very Good Partial Response (VGPR) defined as serum and urine M-component detectable by immunofixation but not on electrophoresis or ≥90% reduction in serum M-component plus urine M-component <100 mg per 24 hours, Partial Response (PR) ≥50% reduction in serum M-component or ≥90% reduction urine M-component or urine M-component <200 mg per 24 hours, Minimal Response (MR) ≥25% reduction in serum or urine M-component, Stable Disease (SD) defined as failure to meet any response criteria, and Progressive Disease (PD) ≥ 25% increase from lowest value reported in serum M-component (absolute ≥0.5 g/dL) and/or urine M-component (absolute ≥200 mg/24 hours).
Time Frame: Disease was assessed for response every cycle on treatment. The maximum number of cycles received was 25.
Population: All participants with measureable disease at baseline and received at least one dose of the study drug were evaluable for response.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase I Dose Level 1 | Phase I Dose Level 2 | Phase I Dose Level 3 | Phase I Dose Level 4 | Phase I Dose Level 5 | Phase I Dose Level 5B | Phase I Dose Level 6 | All Phase II Participants
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 4 | 6 | 3 | 33
Participants
  Complete Response | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
  Very Good Partial Response | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 3
  Partial Response | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 12
  Minimal Response | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 4
  Stable Disease | 3 | 2 | 2 | 0 | 4 | 3 | 2 | 11
  Progressive Disease | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 2

5. Secondary Outcome: Time to Progression (TTP) [Phase II]
Description: TTP estimated using the Kaplan-Meier method is defined as the time from registration to progression based on IMWG criteria or date last known progression-free for those who have not progressed. [Durie BG et al. Leukemia. 2006] Progression (PD): ≥ 25% increase from lowest value reported in serum M-component (absolute increase ≥0.5 g/dL) and/or urine M-component (absolute increase ≥200 mg/24 hours); if appropriate, a ≥25% increase above the lowest level in the difference between involved and uninvolved FLC levels (absolute increase >10 mg/dL); If none of these are measurable then ≥25% increase in bone marrow plasma cell percentage above the lowest response level (absolute ≥10%); Definite development of new bone lesions or soft tissue plasmacytomas OR increase in size of existing
Time Frame: DIsease was assessed to document progression every cycle on treatment and post-treatment every 12 weeks until progression.
Population: All Phase II participants with measureable disease present at baseline and received at least one dose of the study drug were evaluable for TTP.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | All Phase II Participants
Number analyzed (Participants) | 33
Months | 12.6 [5.5 to 23.1]

6. Secondary Outcome: Duration of Response (DOR) [Phase II]
Description: DOR is defined as the time from response to disease progression or death, or date last known progression-free and alive for those who have not progressed or died. DOR was estimated using the Kaplan-Meier method.
Time Frame: DIsease was assessed to document response every cycle on treatment and post-treatment every 12 weeks until progression.
Population: All Phase II participants with measureable disease present at baseline and received at least one dose of the study drug were evaluable for DOR.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | All Phase II Participants
Number analyzed (Participants) | 33
Months | 12.9 [7.8 to 33.3]

ADVERSE EVENTS:
Time Frame: Assessed each treatment cycle from time of first dose and up to day 30 post treatment.
Description: Maximum grade toxicity by type was first calculated. Serius AEs were defined as events with plerixafor, bortezomib and/or dexamethasone (phase II only) treatment-attribution of at least possibly and grade 3 or higher per CTCAE v. 3.0. Other AEs were defined as events with plerixafor, bortezomib and/or dexamethasone (phase II only) treatment-attribution of at least possibly and grades 1 or 2 per CTCAE v. 3.0.
Arm/Group | Phase I Dose Level 1 | Phase I Dose Level 2 | Phase I Dose Level 3 | Phase I Dose Level 4 | Phase I Dose Level 5 | Phase I Dose Level 5B | Phase I Dose Level 6 | All Phase I Participants | All Phase II Participants
Serious Adverse Events (participants affected / at risk) | 1/3 | 1/3 | 0/3 | 2/3 | 2/4 | 2/6 | 0/3 | 8/25 | 14/33
Other Adverse Events (participants affected / at risk) | 3/3 | 3/3 | 3/3 | 3/3 | 4/4 | 6/6 | 3/3 | 25/25 | 33/33
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Phase I Dose Level 1 (N=3) | Phase I Dose Level 2 (N=3) | Phase I Dose Level 3 (N=3) | Phase I Dose Level 4 (N=3) | Phase I Dose Level 5 (N=4) | Phase I Dose Level 5B (N=6) | Phase I Dose Level 6 (N=3) | All Phase I Participants (N=25) | All Phase II Participants (N=33)
Fatigue (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Insomnia (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Anemia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 3 | 3
Lymphocytopenia (Blood and lymphatic system disorders) | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 3 | 3
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 8
Upper airway infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3
Elevated liver function tests (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hyperglycemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hyperlipasemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hyponatremia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hypophosphatemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 2 | 0
Neurologic-other (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Renal/GU-other (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Phase I Dose Level 1 (N=3) | Phase I Dose Level 2 (N=3) | Phase I Dose Level 3 (N=3) | Phase I Dose Level 4 (N=3) | Phase I Dose Level 5 (N=4) | Phase I Dose Level 5B (N=6) | Phase I Dose Level 6 (N=3) | All Phase I Participants (N=25) | All Phase II Participants (N=33)
Allergic reaction (Immune system disorders) | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 3 | 1
Allergic rhinitis (Immune system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Allergy-other (Immune system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Hearing w/o audiogr not in monitor prg (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hematologic-other (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Cardiac-other (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3
Hypertension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3
Hypotension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Constitutional- other (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3
Fatigue (General disorders) | 3 | 3 | 1 | 2 | 4 | 5 | 3 | 21 | 18
Fever w/o neutropenia (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 3
Insomnia (Psychiatric disorders) | 2 | 1 | 0 | 0 | 1 | 1 | 2 | 7 | 13
Rigors/chills (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Sweating (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 2
Weight gain (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Weight loss (Investigations) | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 3 | 1
Bruising (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 2
Erythema multiforme (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Induration/fibrosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Injection site reaction (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 1
Pruritus/itching (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 2 | 1
Rash/desquamation (Skin and subcutaneous tissue disorders) | 2 | 0 | 0 | 1 | 2 | 1 | 0 | 6 | 1
Rash: acne/acneiform (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Endocrine-other (Endocrine disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hot flashes (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1
Anorexia (Metabolism and nutrition disorders) | 2 | 2 | 0 | 0 | 0 | 0 | 0 | 4 | 5
Constipation (Gastrointestinal disorders) | 2 | 0 | 0 | 0 | 0 | 1 | 1 | 4 | 11
Dehydration (Metabolism and nutrition disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 3
Diarrhea (Gastrointestinal disorders) | 1 | 1 | 2 | 2 | 4 | 4 | 2 | 16 | 21
Distention/bloating- abdominal (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 2 | 1
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 3
Flatulence (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
GI-other (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 4
Muco/stomatitis (symptom) oral cavity (Gastrointestinal disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 2 | 0
Nausea (Gastrointestinal disorders) | 1 | 3 | 1 | 2 | 2 | 2 | 1 | 12 | 11
Obstruction- small bowel NOS (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Taste disturbance (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Ulcer- gastric (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 3 | 2
Hemorrhage-other (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Nose- hemorrhage (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Anemia (Blood and lymphatic system disorders) | 3 | 2 | 0 | 1 | 1 | 4 | 0 | 11 | 13
Leukocytopenia (Blood and lymphatic system disorders) | 1 | 2 | 0 | 0 | 2 | 0 | 1 | 6 | 4
Lymphocytopenia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 1 | 1 | 1 | 4 | 2
Neutropenia (Blood and lymphatic system disorders) | 1 | 1 | 0 | 0 | 1 | 0 | 1 | 4 | 2
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 3 | 0 | 1 | 0 | 3 | 1 | 9 | 6
Infection Gr0-2 neut- eye NOS (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Infection Gr0-2 neut- lip/perioral (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Infection Gr0-2 neut- middle ear (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Infection Gr0-2 neut- skin (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Infection Gr0-2 neut- upper airway (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 4
Infection w/ gr3-4 neut- colon (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Infection w/ unk ANC sinus (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Infection w/ unk ANC urinary tract NOS (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Infection-other (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3
Upper airway infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 4
Edema head and neck (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Edema limb (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 2 | 4
Alkaline phosphatase (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 3
Bicarbonate (Investigations) | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 3 | 2
Bilirubin (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2
Creatinine (Investigations) | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 3 | 5
Elevated liver function tests (Investigations) | 2 | 0 | 1 | 0 | 0 | 0 | 0 | 3 | 4
Hypercalcemia (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Hypercholesterolemia (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hyperglycemia (Metabolism and nutrition disorders) | 2 | 2 | 0 | 0 | 1 | 1 | 0 | 6 | 6
Hyperkalemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Hypoalbuminemia (Metabolism and nutrition disorders) | 2 | 1 | 0 | 0 | 0 | 2 | 1 | 6 | 8
Hypocalcemia (Metabolism and nutrition disorders) | 3 | 1 | 0 | 0 | 0 | 1 | 2 | 7 | 5
Hypoglycemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Hypokalemia (Metabolism and nutrition disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 1 | 3 | 2
Hypomagnesemia (Metabolism and nutrition disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 3
Hyponatremia (Metabolism and nutrition disorders) | 3 | 1 | 0 | 0 | 0 | 0 | 0 | 4 | 4
Hypophosphatemia (Metabolism and nutrition disorders) | 2 | 2 | 2 | 2 | 1 | 0 | 1 | 10 | 5
Metabolic/Laboratory-other (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 6
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Fracture (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Musculoskeletal/soft tissue-other (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3
Nonneuropathic generalized weakness (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 0 | 1 | 0 | 1 | 4 | 5
Agitation (Psychiatric disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 3 | 0
Anxiety (Psychiatric disorders) | 0 | 1 | 1 | 1 | 0 | 0 | 1 | 4 | 3
Confusion (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 0
Depression (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 2
Dizziness (Nervous system disorders) | 1 | 0 | 0 | 2 | 1 | 1 | 0 | 5 | 4
Extrapyramidal movement (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 2 | 0
Mental status (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Neurologic-other (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Neuropathy CN IV down/in eye move (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Neuropathy CN XII tongue (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Neuropathy, sensory (Nervous system disorders) | 3 | 2 | 2 | 1 | 1 | 1 | 2 | 12 | 19
Neuropathy-motor (Nervous system disorders) | 0 | 0 | 0 | 1 | 1 | 2 | 0 | 4 | 0
Personality (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Psychosis (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 2 | 0
Tremor (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Double vision (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Eyelid dysfunction (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 1
Ocular-other (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 2
Vision-blurred (Eye disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Abdomen- pain (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 1 | 1 | 0 | 4 | 1
Anus- pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Back- pain (Musculoskeletal and connective tissue disorders) | 3 | 0 | 0 | 0 | 2 | 2 | 0 | 7 | 10
Bone- pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 1 | 1 | 2 | 1 | 0 | 7 | 2
Chest wall- pain (Musculoskeletal and connective tissue disorders) | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 1
Dental/teeth/peridontal- pain (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Extremity-limb- pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 2 | 1
Eye- pain (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Head/headache (Nervous system disorders) | 0 | 2 | 0 | 2 | 1 | 1 | 0 | 6 | 6
Joint- pain (Musculoskeletal and connective tissue disorders) | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 5
Larynx- pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Middle ear- pain (Ear and labyrinth disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Muscle- pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1 | 1 | 0 | 1 | 4 | 2
Neck- pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 2 | 1
Neuropathic- pain (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Pain-other (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 5
Testicle- pain (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 3 | 3
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 6
Incontinence urinary (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1
Renal/GU-other (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1
Urinary frequency/urgency (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Intra-op injury Other (Specify) (Surgical and medical procedures) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No